CLINICAL TRIAL: NCT00879151
Title: Treatment of Bulimic Adolescents
Brief Title: Study of Treatment for Adolescents With Bulimia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Principal Investigator, James Dale Lock, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-02272009-1878; eProtocol Number 132056
Record Dates: First submitted 2009-04-07; First posted 2009-04-09 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Bulimia
MeSH Terms: conditions — Bulimia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Psychotherapy (Experimental): Patients are randomized to one of three different types of psychotherapy: Cognitive-Behavioral Therapy for adolescents, Family-Based Therapy for Bulimia Nervosa, and Supportive Psychotherapy. All treatments consist of 18 sessions over a period of approximately 6 months.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Adolescents; Behavioral: Supportive Psychotherapy; Behavioral: Family Based Therapy for Bulimia Nervosa

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Adolescents — The therapist will work with the adolescent to understand triggers to binge eating and purging, such as thoughts, feelings, and interpersonal difficulties. Also, establishing regular eating patterns and eliminating medically harmful behaviors associated with the eating disorder is a primary goal.
Behavioral: Supportive Psychotherapy — SPT focuses on having the patient build a relationship with the therapist and explore their unique individual needs within the context of their life and the experience of having an eating disorder.
Behavioral: Family Based Therapy for Bulimia Nervosa — FBT helps parents to take an active role in guiding their child through eating disorder treatment. In this therapy, the parents are supported in helping their child stop bingeing, purging and engaging in other harmful weight-control behaviors. The way in which the eating disorder has impacted the family and the adolescent's development is also explored.

SUMMARY:
In the face of scant literature on the subject, the investigators aim to more clearly identify effective treatments for adolescent bulimia nervosa (BN) through a treatment study comparing two current treatments (Cognitive Behavioral Therapy for Adolescents, CBT-A and Family Based Therapy for Bulimia Nervosa, FBT-BN) for the disorder in comparison with a non-specific therapy, Supportive Psychotherapy for Adolescent Bulimia (SPT). Additionally, the investigators hope to provide clinicians with information on treatment efficacy, variables that might influence outcome, and processes that may affect treatment efficacy that will guide them in their efforts to treat adolescent BN.

DETAILED DESCRIPTION:
BN is a serious disorder that is characterized by extreme concerns about body weight and shape, dieting, and the disinhibited eating behaviors of binging and purging. There are no published randomized clinical trials of psychotherapy treatment for Bulimia Nervosa in adolescents although it often onsets in this age group. There is evidence that some treatments are effective, but none has been empirically tested. Because Bulimia Nervosa is a serious medical and psychiatric illness it is important to learn efficacious ways to treat this disorder, especially in its early stages. Treatments used in this study are the best known treatments for adults with Bulimia Nervosa. The investigators hope to learn which of two previously studied treatments might be superior to the other, in an effort to guide clinicians in treatment choices. Successfully treating the disorder early on (even in those adolescents with partial BN, characterized by binge eating and purging at least one time per week over a 6 month period) may reduce the number of cases requiring treatment during adulthood, leading to possible reduction in severity of associated psychopathology and lower costs, as well as enable individuals to lead more productive lives.

Given the neglect of adolescent BN in the research literature and the need for information to guide the clinical treatment of this disorder, this study's primary aim is to compare the efficacy of CBT-A to FBT-BN in decreasing binge eating and purging episodes in adolescents with BN and partial BN (defined as binge eating and purging at least one time per week for the past six months).

Participation in this study will last 1 and a half years and will consist of 6 months of treatment and a follow-up session at 6 and 12 months post-treatment. All participants will first undergo baseline assessments, which include interviews and questionnaires about psychological history and BN symptoms, and an Eating Disorder Examination (EDE) interview. All treatment assignments consist of 18 sessions of therapy over the course of 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be adolescents living with at least one of their parents and between the ages of 12 and 18 years of age with a DSM IV diagnosis of BN or partial BN (binge eating and purging at least one time per week over a six month period).
2. Males meeting inclusion criteria will also be entered into the study. They must have age-adjusted BMI greater than 17.5, or ideal body weight (IBW) > 85%.
3. Family, for the purposes of this study, includes members of the subject's household, including at least one parent or adult guardian. Single parent families, divorced families, step-parents, and other types of families will be allowed to enter the study.

Exclusion Criteria:

1. psychotic illness or other mental illness requiring hospitalization; bipolar I disorder, depression with active suicidal thoughts and behavior;
2. associated physical illness that necessitates hospitalization;
3. current dependence on drugs or alcohol;
4. current diagnosis of anorexia nervosa or weight less that 85% IBW;
5. physical conditions (e.g. diabetes mellitus, pregnancy) known to influence eating or weight;
6. currently taking medication for co-morbid conditions for less than 2-months;
7. currently taking medications that may induce weight loss, e.g., appetite suppressants such as sibutramine, phentermine, and xenical, unless the participant is willing to withdraw from such medications;
8. currently taking medications for symptoms of BN and unwilling to discontinue these prior to initiating treatment in the study
9. previous CBT or FBT treatment for BN
10. married subjects
11. emancipated minors
12. family members will be excluded from engaging in treatment for the following reasons:

    * Current or history of sexual or physical abuse of the patient by family members. Perpetrators of the abuse will be excluded from treatment. Should sexual or physical abuse by a family member occur during the course of treatment, perpetrators will be excluded from ongoing treatment.
    * Substance dependence, psychosis, or severe medical illness that would limit full participation in therapy, or that might put the family member at risk for worsening of their condition during treatment. The decision whether or not to allow these individuals to continue to participate in treatment will be made by the therapist in consultation with the treatment supervisor.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2009-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Binge and purge frequency as assessed by the Eating Disorder Examination (EDE) | End of Treatment

SECONDARY OUTCOMES:
Changes in the subscale scores of the EDE | End of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: James D Lock, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - University of Chicago, Chicago, Illinois

REFERENCES:
- [Derived] Gorrell S, Kinasz K, Hail L, Bruett L, Forsberg S, Lock J, Le Grange D. Rituals and preoccupations associated with bulimia nervosa in adolescents: Does motivation to change matter? Eur Eat Disord Rev. 2019 May;27(3):323-328. doi: 10.1002/erv.2664. Epub 2019 Feb 7. PMID 30734406
- [Derived] Valenzuela F, Lock J, Le Grange D, Bohon C. Comorbid depressive symptoms and self-esteem improve after either cognitive-behavioural therapy or family-based treatment for adolescent bulimia nervosa. Eur Eat Disord Rev. 2018 May;26(3):253-258. doi: 10.1002/erv.2582. Epub 2018 Feb 15. PMID 29446174
- [Derived] Le Grange D, Lock J, Agras WS, Bryson SW, Jo B. Randomized Clinical Trial of Family-Based Treatment and Cognitive-Behavioral Therapy for Adolescent Bulimia Nervosa. J Am Acad Child Adolesc Psychiatry. 2015 Nov;54(11):886-94.e2. doi: 10.1016/j.jaac.2015.08.008. Epub 2015 Sep 2. PMID 26506579
- [Derived] Darcy AM, Fitzpatrick KK, Manasse SM, Datta N, Klabunde M, Colborn D, Aspen V, Stiles-Shields C, Labuschagne Z, Le Grange D, Lock J. Central coherence in adolescents with bulimia nervosa spectrum eating disorders. Int J Eat Disord. 2015 Jul;48(5):487-93. doi: 10.1002/eat.22340. Epub 2014 Aug 22. PMID 25146149
- [Derived] Darcy AM, Fitzpatrick KK, Colborn D, Manasse S, Datta N, Aspen V, Shields CS, Le Grange D, Lock J. Set-shifting among adolescents with bulimic spectrum eating disorders. Psychosom Med. 2012 Oct;74(8):869-72. doi: 10.1097/PSY.0b013e31826af636. Epub 2012 Sep 21. PMID 23001391